CLINICAL TRIAL: NCT06590428
Title: Therapeutic Drug Monitoring for Linezolid in the Treatment of Rifampin-resistant Tuberculosis
Acronym: THERMOL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: University of Cape Town (Other); St George's, University of London (Other); Emory University (Other); National Department of Health, South Africa (Unknown); Columbia University (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-16182; R01AI184416 (NIH)
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Rifampin-resistant Tuberculosis; Drug-resistant Tuberculosis
Keywords: HIV Status; Therapeutic Drug Monitoring; anti-Tuberculosis activity; Linezolid
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant | interventions — Linezolid

STUDY DESIGN:
Intervention Model Description: 1:1 randomization.
  Participants will receive 600mg daily dose of oral LZD for Rifampicin-resistant tuberculosis (RR-TB) as part of standard of care for both arms. This dosage may be reduced to 300mg daily based on the plasma trough concentration obtained from the first pharmacokinetic (PK) specimen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Therapeutic Drug Monitoring (TDM) (Other): Participants in the TDM arm will have their linezolid dose reduced if their trough concentration is greater than 2.5 mg/L
  Interventions: Other: Therapeutic Drug Monitoring for Linezolid
- Standard of Care (SOC) (No Intervention): Participants in the SOC arm will have their linezolid adjusted or held if they develop clinical adverse events.

INTERVENTIONS:
Other: Therapeutic Drug Monitoring for Linezolid — TDM with dose adjustment for trough concentration >2.5 mg/L LZD
  Arms: Therapeutic Drug Monitoring (TDM)

SUMMARY:
This study is a two-arm, pragmatic, open-label, randomized clinical trial to determine the efficacy of Therapeutic Drug Monitoring (TDM) in preventing premature discontinuation of Linezolid (LZD) in participants with Rifampicin-resistant tuberculosis (RR-TB). Following the initiation of treatment, participants will be monitored throughout the approximate 6-month duration of RR-TB therapy.

DETAILED DESCRIPTION:
Drug-resistant tuberculosis (TB) is a major global epidemic and poses a particular threat to HIV-infected individuals. With limited effective drugs available for treatment, multidrug-, and extensively drug-resistant TB carry a high mortality rate and threaten global TB and HIV control efforts.

New and repurposed medications have recently been found to improve survival and cure rates. Linezolid-a drug initially developed for the treatment of Gram-positive infections-has considerable anti-TB activity and has been at the center of this treatment revolution. Since 2018, WHO has recommended that all multi DR/rifampicin-resistant (MDR) and extensively drug-resistant tuberculosis (XDR) tuberculosis treatment regimens include linezolid. When given long-term, however, linezolid-associated toxicity-particularly myelosuppression and peripheral neuropathy-is very common, affecting 50-80% of patients and often requiring a temporary or permanent discontinuation of therapy. Such interruptions put patients at risk of treatment failure and the emergence of additional resistance to linezolid or one of the other drugs in the regimen. As linezolid use continues to increase worldwide, such resistance could become widespread, squandering a valuable medication. Previously conducted research has shown that linezolid toxicities are associated with trough plasma concentration and that the drug has considerable inter-individual variability. The investigator team, therefore, hypothesize that therapeutic drug monitoring (TDM) could identify those with higher linezolid concentrations and permit pre-emptive dose reductions that could avert drug toxicity and premature discontinuation.

This study will take place at the Nkqubela TB Specialist Hospital in East London, South Africa. TB diagnosis and initial treatment regimen will be determined by the hospital clinical team, per local guidelines. Following enrollment, participants will be randomized after enrollment to either undergo a therapeutic drug monitoring (TDM) strategy for LZD, or standard of care (SOC). Participants in both arms will have a trough plasma linezolid concentration drawn approximately one week after enrollment (within one month of TB treatment initiation). The PK specimens collected from TDM arm participants will be analyzed by University of Cape Town lab staff. The PK specimens collected from SOC participants will be stored for future analysis.

Standard treatment for RR-TB in South Africa includes 6 months of therapy, including linezolid 600 mg daily for duration of treatment. Those in the TDM arm whose concentration is above a set threshold (2.5 mg/L) will have their LZD dose reduced to 300mg daily, while those in the SOC arm will receive routine monitoring alone. All participants will be screened monthly for hematologic and neurologic toxicity. Hospital and clinic providers will manage all treatment other than the TDM-guided linezolid dose reduction. If participants in either the SOC or TDM arm experience linezolid toxicity, hospital and clinic providers may choose to temporarily or permanently discontinue linezolid, regardless of any prior TDM-guided dose reduction, in accordance with South African national guidelines.

Aim 1 (Primary Outcome Measure of this study) and Aim 2 (the first Secondary Outcome Measure) are described in the Outcome Measures section. For Aim 3, population PK modeling will be used to explore the complex relationship between linezolid pharmacokinetic parameters and the trajectory of toxicities over time. It will also be determined as to whether those whose dose is lowered still meet exposure targets for drug efficacy. South Africa has among the highest global burden of drug-resistant TB and HIV and has led the world in the rollout of new RR-TB drugs and regimens. The aims of this study will answer fundamental questions about LZD pharmacology that will directly inform its use in South Africa and worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patient > 18 years of age
* Microbiological confirmation of rifampicin-resistant tuberculosis (e.g., phenotypic drug susceptibility testing, GeneXpert MTB/RIF™). Participants may have resistance to additional medications as well - i.e., MDR and XDR TB - but must have resistance to at least rifampin
* Initiated on a RR-TB treatment regimen containing linezolid, no more than 14 days prior to enrollment
* HIV status is known

  * Both HIV-positive and HIV-negative individuals are eligible
  * If an individual reports unknown HIV results, they must consent to HIV testing at time of enrollment to confirm status. If they decline to be tested, they are not eligible for the study
  * If an individual declines to share his or her HIV status, they are not eligible for the study. Patients reporting unknown HIV status will be required to have had confirmatory testing within 6 months of study screening

Exclusion Criteria:

* Current unstable or uncontrolled major medical comorbidity that would interfere with subject's ability to participate in the study
* Pregnant at time of screening
* Initial linezolid dose < 600mg daily

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Discontinuation of Linezolid or non-TDM guided dose reduction | Within 6 months after initiation of LZD therapy
  Linezolid (LZD) discontinuation for any cause along with non-TDM-guided LZD dose reduction will be assessed. The number of participants who discontinue LZD (defined as an interruption > 2 weeks in duration), including self-discontinuation by the patient or a decision by the provider to temporarily or permanently discontinue LZD, OR have a non-TDM-guided dose-reduction in response to an adverse event, will be summarized by study arm using basic descriptive statistics.

SECONDARY OUTCOMES:
Evidence of Linezolid Toxicity | Within 6 months after initiation of LZD therapy
  Evidence of Linezolid (LZD) toxicity will be evaluated by the number of participants who experience Grade 3 or Grade 4 hematologic or neurologic adverse events associated with LZD toxicity. LZD-associated Grade 3 or Grade 4 events, documented at any time point up to 6 months, will be summarized by adverse event type and frequency for each study arm.
Unsuccessful final Tuberculosis (TB) end-of-treatment outcome | After 6 months, and up to 12 months after initiation of LZD therapy
  Unsuccessful final TB treatment outcome is defined as either treatment failure, death, or participant lost to follow-up, as per World Health Organization (WHO) definitions, defined below. End-of-treatment TB outcomes will be captured for all study participants. The number of participants with unsuccessful final TB treatment outcomes will be summarized by study arm using basic descriptive statistics. TB treatment outcomes will be assessed at the end of 6 months of treatment; however, if treatment is extended for any reason, medical records will be reviewed 12 months after treatment initiation to capture a final TB treatment outcome.
  Treatment failure: The patient's treatment was terminated or they needed to permanently change their regimen due to a lack of response to treatment, adverse drug reaction, or increased drug resistance.
  Lost to follow-up: The patient stopped taking their medication for two or more months in a row after registering.
  Death: The patient died
Emergence of new phenotypic resistance to Linezolid | Within 6 months after initiation of LZD therapy
  The percentage of participants in each arm who develop phenotypic Linezolid (LZD) resistance will be assessed. Participants who experience treatment failure and remain sputum culture-positive after 4 months, will have a sputum sample collected for additional drug-resistance testing. Results of any isolates which undergo such resistance testing will be reviewed to identify anyone with treatment-emergent linezolid resistance. Additionally, during follow-up visits, participants will be directly assessed for development of LZD resistance. The percentage of participants who develop phenotypic resistance to LZD, as determined by either of these methods, will be summarized by study arm using basic descriptive statistics

CONTACTS AND LOCATIONS:
Overall Officials: James CM Brust, MD, Principal Investigator — Albert Einstein College of Medicine; Gary Maartens, MBChB, Principal Investigator — University of Cape Town
Locations (1):
- Nkqubela TB Specialist Hospital, East London, Eastern Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization. Global Tuberculosis Report 2022. Geneva.
- [Background] Shah NS, Wright A, Bai GH, Barrera L, Boulahbal F, Martin-Casabona N, Drobniewski F, Gilpin C, Havelkova M, Lepe R, Lumb R, Metchock B, Portaels F, Rodrigues MF, Rusch-Gerdes S, Van Deun A, Vincent V, Laserson K, Wells C, Cegielski JP. Worldwide emergence of extensively drug-resistant tuberculosis. Emerg Infect Dis. 2007 Mar;13(3):380-7. doi: 10.3201/eid1303.061400. PMID 17552090
- [Background] Migliori GB, Sotgiu G, Gandhi NR, Falzon D, DeRiemer K, Centis R, Hollm-Delgado MG, Palmero D, Perez-Guzman C, Vargas MH, D'Ambrosio L, Spanevello A, Bauer M, Chan ED, Schaaf HS, Keshavjee S, Holtz TH, Menzies D; "The Collaborative Group for Meta-Analysis of Individual Patient Data in MDR-TB". Drug resistance beyond extensively drug-resistant tuberculosis: individual patient data meta-analysis. Eur Respir J. 2013 Jul;42(1):169-179. doi: 10.1183/09031936.00136312. Epub 2012 Oct 11. PMID 23060633
- [Background] Centers for Disease Control and Prevention (CDC). Emergence of Mycobacterium tuberculosis with extensive resistance to second-line drugs--worldwide, 2000-2004. MMWR Morb Mortal Wkly Rep. 2006 Mar 24;55(11):301-5. PMID 16557213
- [Background] Gandhi NR, Shah NS, Andrews JR, Vella V, Moll AP, Scott M, Weissman D, Marra C, Lalloo UG, Friedland GH; Tugela Ferry Care and Research (TF CARES) Collaboration. HIV coinfection in multidrug- and extensively drug-resistant tuberculosis results in high early mortality. Am J Respir Crit Care Med. 2010 Jan 1;181(1):80-6. doi: 10.1164/rccm.200907-0989OC. Epub 2009 Oct 15. PMID 19833824
- [Background] Migliori GB, Besozzi G, Girardi E, Kliiman K, Lange C, Toungoussova OS, Ferrara G, Cirillo DM, Gori A, Matteelli A, Spanevello A, Codecasa LR, Raviglione MC; SMIRA/TBNET Study Group. Clinical and operational value of the extensively drug-resistant tuberculosis definition. Eur Respir J. 2007 Oct;30(4):623-6. doi: 10.1183/09031936.00077307. Epub 2007 Aug 9. PMID 17690121
- [Background] Shah NS, Pratt R, Armstrong L, Robison V, Castro KG, Cegielski JP. Extensively drug-resistant tuberculosis in the United States, 1993-2007. JAMA. 2008 Nov 12;300(18):2153-60. doi: 10.1001/jama.300.18.2153. PMID 19001626
- [Background] Gandhi NR, Moll A, Sturm AW, Pawinski R, Govender T, Lalloo U, Zeller K, Andrews J, Friedland G. Extensively drug-resistant tuberculosis as a cause of death in patients co-infected with tuberculosis and HIV in a rural area of South Africa. Lancet. 2006 Nov 4;368(9547):1575-80. doi: 10.1016/S0140-6736(06)69573-1. PMID 17084757
- [Background] Pietersen E, Ignatius E, Streicher EM, Mastrapa B, Padanilam X, Pooran A, Badri M, Lesosky M, van Helden P, Sirgel FA, Warren R, Dheda K. Long-term outcomes of patients with extensively drug-resistant tuberculosis in South Africa: a cohort study. Lancet. 2014 Apr 5;383(9924):1230-9. doi: 10.1016/S0140-6736(13)62675-6. Epub 2014 Jan 17. PMID 24439237
- [Background] Schnippel K, Ndjeka N, Maartens G, Meintjes G, Master I, Ismail N, Hughes J, Ferreira H, Padanilam X, Romero R, Te Riele J, Conradie F. Effect of bedaquiline on mortality in South African patients with drug-resistant tuberculosis: a retrospective cohort study. Lancet Respir Med. 2018 Sep;6(9):699-706. doi: 10.1016/S2213-2600(18)30235-2. Epub 2018 Jul 11. PMID 30001994
- [Background] Collaborative Group for the Meta-Analysis of Individual Patient Data in MDR-TB treatment-2017; Ahmad N, Ahuja SD, Akkerman OW, Alffenaar JC, Anderson LF, Baghaei P, Bang D, Barry PM, Bastos ML, Behera D, Benedetti A, Bisson GP, Boeree MJ, Bonnet M, Brode SK, Brust JCM, Cai Y, Caumes E, Cegielski JP, Centis R, Chan PC, Chan ED, Chang KC, Charles M, Cirule A, Dalcolmo MP, D'Ambrosio L, de Vries G, Dheda K, Esmail A, Flood J, Fox GJ, Frechet-Jachym M, Fregona G, Gayoso R, Gegia M, Gler MT, Gu S, Guglielmetti L, Holtz TH, Hughes J, Isaakidis P, Jarlsberg L, Kempker RR, Keshavjee S, Khan FA, Kipiani M, Koenig SP, Koh WJ, Kritski A, Kuksa L, Kvasnovsky CL, Kwak N, Lan Z, Lange C, Laniado-Laborin R, Lee M, Leimane V, Leung CC, Leung EC, Li PZ, Lowenthal P, Maciel EL, Marks SM, Mase S, Mbuagbaw L, Migliori GB, Milanov V, Miller AC, Mitnick CD, Modongo C, Mohr E, Monedero I, Nahid P, Ndjeka N, O'Donnell MR, Padayatchi N, Palmero D, Pape JW, Podewils LJ, Reynolds I, Riekstina V, Robert J, Rodriguez M, Seaworth B, Seung KJ, Schnippel K, Shim TS, Singla R, Smith SE, Sotgiu G, Sukhbaatar G, Tabarsi P, Tiberi S, Trajman A, Trieu L, Udwadia ZF, van der Werf TS, Veziris N, Viiklepp P, Vilbrun SC, Walsh K, Westenhouse J, Yew WW, Yim JJ, Zetola NM, Zignol M, Menzies D. Treatment correlates of successful outcomes in pulmonary multidrug-resistant tuberculosis: an individual patient data meta-analysis. Lancet. 2018 Sep 8;392(10150):821-834. doi: 10.1016/S0140-6736(18)31644-1. PMID 30215381
- [Background] Conradie F, Diacon A, Howell P, et al. Sustained high rate of successful treatment outcomes: Interim results of 75 patients in the Nix-TB clinical study of pretomanid, bedaquiline and linezolid. 49th Union World Conference on Lung Health The Hague, Netherlands 24-27 October 2018 Abstract OA03-213-25.
- [Background] Diacon AH, De Jager VR, Dawson R, Narunsky K, Vanker N, Burger DA, Everitt D, Pappas F, Nedelman J, Mendel CM. Fourteen-Day Bactericidal Activity, Safety, and Pharmacokinetics of Linezolid in Adults with Drug-Sensitive Pulmonary Tuberculosis. Antimicrob Agents Chemother. 2020 Mar 24;64(4):e02012-19. doi: 10.1128/AAC.02012-19. Print 2020 Mar 24. PMID 31988102
- [Background] Zurenko GE, Yagi BH, Schaadt RD, Allison JW, Kilburn JO, Glickman SE, Hutchinson DK, Barbachyn MR, Brickner SJ. In vitro activities of U-100592 and U-100766, novel oxazolidinone antibacterial agents. Antimicrob Agents Chemother. 1996 Apr;40(4):839-45. doi: 10.1128/AAC.40.4.839. PMID 8849237
- [Background] Cynamon MH, Klemens SP, Sharpe CA, Chase S. Activities of several novel oxazolidinones against Mycobacterium tuberculosis in a murine model. Antimicrob Agents Chemother. 1999 May;43(5):1189-91. doi: 10.1128/AAC.43.5.1189. PMID 10223934
- [Background] Lee M, Lee J, Carroll MW, Choi H, Min S, Song T, Via LE, Goldfeder LC, Kang E, Jin B, Park H, Kwak H, Kim H, Jeon HS, Jeong I, Joh JS, Chen RY, Olivier KN, Shaw PA, Follmann D, Song SD, Lee JK, Lee D, Kim CT, Dartois V, Park SK, Cho SN, Barry CE 3rd. Linezolid for treatment of chronic extensively drug-resistant tuberculosis. N Engl J Med. 2012 Oct 18;367(16):1508-18. doi: 10.1056/NEJMoa1201964. PMID 23075177
- [Background] Conradie F, Diacon AH, Ngubane N, Howell P, Everitt D, Crook AM, Mendel CM, Egizi E, Moreira J, Timm J, McHugh TD, Wills GH, Bateson A, Hunt R, Van Niekerk C, Li M, Olugbosi M, Spigelman M; Nix-TB Trial Team. Treatment of Highly Drug-Resistant Pulmonary Tuberculosis. N Engl J Med. 2020 Mar 5;382(10):893-902. doi: 10.1056/NEJMoa1901814. PMID 32130813
- [Background] Conradie F, Bagdasaryan TR, Borisov S, Howell P, Mikiashvili L, Ngubane N, Samoilova A, Skornykova S, Tudor E, Variava E, Yablonskiy P, Everitt D, Wills GH, Sun E, Olugbosi M, Egizi E, Li M, Holsta A, Timm J, Bateson A, Crook AM, Fabiane SM, Hunt R, McHugh TD, Tweed CD, Foraida S, Mendel CM, Spigelman M; ZeNix Trial Team. Bedaquiline-Pretomanid-Linezolid Regimens for Drug-Resistant Tuberculosis. N Engl J Med. 2022 Sep 1;387(9):810-823. doi: 10.1056/NEJMoa2119430. PMID 36053506
- [Background] Nyang'wa BT, Berry C, Kazounis E, Motta I, Parpieva N, Tigay Z, Solodovnikova V, Liverko I, Moodliar R, Dodd M, Ngubane N, Rassool M, McHugh TD, Spigelman M, Moore DAJ, Ritmeijer K, du Cros P, Fielding K; TB-PRACTECAL Study Collaborators. A 24-Week, All-Oral Regimen for Rifampin-Resistant Tuberculosis. N Engl J Med. 2022 Dec 22;387(25):2331-2343. doi: 10.1056/NEJMoa2117166. PMID 36546625
- [Background] World Health Organization. Treatment guidelines for multidrug- and rifampicin-resistant tuberculosis: 2018 update; Pre-final text; WHO/CDS/TB/2018.15 Geneva.
- [Background] Department of Health South Africa. Clinical Management of Rifampin-Resistant Tuberculosis: Updated Clinical Reference Guide. 2023.
- [Background] WHO consolidated guidelines on tuberculosis: Module 4: Treatment - Drug-resistant tuberculosis treatment [Internet]. Geneva: World Health Organization; 2020. Available from http://www.ncbi.nlm.nih.gov/books/NBK558570/ PMID 32603040
- [Background] World Health Organization. The END TB Strategy. WHO/HTM/TB/201519; Geneva, Switzerland 2015.
- [Background] Fauci AS, Eisinger RW. Reimagining the Research Approach to Tuberculosisdagger. Am J Trop Med Hyg. 2018 Mar;98(3):650-652. doi: 10.4269/ajtmh.17-0999. Epub 2018 Jan 11. PMID 29363452
- [Background] De Vriese AS, Coster RV, Smet J, Seneca S, Lovering A, Van Haute LL, Vanopdenbosch LJ, Martin JJ, Groote CC, Vandecasteele S, Boelaert JR. Linezolid-induced inhibition of mitochondrial protein synthesis. Clin Infect Dis. 2006 Apr 15;42(8):1111-7. doi: 10.1086/501356. Epub 2006 Mar 13. PMID 16575728
- [Background] Zyvox [package insert]; https://www.accessdata.fda.gov/drugsatfda_docs/label/2014/021130s032,021131s026,021132s031lbl.pdf (accessed Sep 10, 2023).
- [Background] Sotgiu G, Centis R, D'Ambrosio L, Alffenaar JW, Anger HA, Caminero JA, Castiglia P, De Lorenzo S, Ferrara G, Koh WJ, Schecter GF, Shim TS, Singla R, Skrahina A, Spanevello A, Udwadia ZF, Villar M, Zampogna E, Zellweger JP, Zumla A, Migliori GB. Efficacy, safety and tolerability of linezolid containing regimens in treating MDR-TB and XDR-TB: systematic review and meta-analysis. Eur Respir J. 2012 Dec;40(6):1430-42. doi: 10.1183/09031936.00022912. Epub 2012 Apr 10. PMID 22496332
- [Background] Cox H, Ford N. Linezolid for the treatment of complicated drug-resistant tuberculosis: a systematic review and meta-analysis. Int J Tuberc Lung Dis. 2012 Apr;16(4):447-54. doi: 10.5588/ijtld.11.0451. PMID 22325685
- [Background] Zhang X, Falagas ME, Vardakas KZ, Wang R, Qin R, Wang J, Liu Y. Systematic review and meta-analysis of the efficacy and safety of therapy with linezolid containing regimens in the treatment of multidrug-resistant and extensively drug-resistant tuberculosis. J Thorac Dis. 2015 Apr;7(4):603-15. doi: 10.3978/j.issn.2072-1439.2015.03.10. PMID 25973226
- [Background] Kwon YS, Jang JG, Lee J, Choi KJ, Park JE. Risk factors for peripheral neuropathy in patients on linezolid-containing regimens for drug-resistant TB. Int J Tuberc Lung Dis. 2023 Mar 1;27(3):232-234. doi: 10.5588/ijtld.22.0423. No abstract available. PMID 36855040
- [Background] Padmapriyadarsini C, Solanki R, Jeyakumar SM, Bhatnagar A, Muthuvijaylaksmi M, Jeyadeepa B, Reddy D, Shah P, Sridhar R, Vohra V, Bhui NK. Linezolid Pharmacokinetics and Its Association with Adverse Drug Reactions in Patients with Drug-Resistant Pulmonary Tuberculosis. Antibiotics (Basel). 2023 Apr 6;12(4):714. doi: 10.3390/antibiotics12040714. PMID 37107075
- [Background] Wasserman S, Meintjes G, Maartens G. Linezolid in the treatment of drug-resistant tuberculosis: the challenge of its narrow therapeutic index. Expert Rev Anti Infect Ther. 2016 Oct;14(10):901-15. doi: 10.1080/14787210.2016.1225498. Epub 2016 Aug 27. PMID 27532292
- [Background] Cattaneo D, Marriott DJ, Gervasoni C. Hematological toxicities associated with linezolid therapy in adults: key findings and clinical considerations. Expert Rev Clin Pharmacol. 2023 Mar;16(3):219-230. doi: 10.1080/17512433.2023.2181160. Epub 2023 Feb 21. PMID 36787631
- [Background] Cattaneo D, Baldelli S, Cerea M, Landonio S, Meraviglia P, Simioni E, Cozzi V, Fucile S, Gazzaniga A, Clementi E, Galli M, Rizzardini G, Gervasoni C. Comparison of the in vivo pharmacokinetics and in vitro dissolution of raltegravir in HIV patients receiving the drug by swallowing or by chewing. Antimicrob Agents Chemother. 2012 Dec;56(12):6132-6. doi: 10.1128/AAC.00942-12. Epub 2012 Sep 10. PMID 22964253
- [Background] Zhang H, He Y, Davies Forsman L, Paues J, Werngren J, Niward K, Schon T, Bruchfeld J, Alffenaar JW, Hu Y. Population pharmacokinetics and dose evaluations of linezolid in the treatment of multidrug-resistant tuberculosis. Front Pharmacol. 2023 Jan 9;13:1032674. doi: 10.3389/fphar.2022.1032674. eCollection 2022. PMID 36699070
- [Background] Alghamdi WA, Al-Shaer MH, An G, Alsultan A, Kipiani M, Barbakadze K, Mikiashvili L, Ashkin D, Griffith DE, Cegielski JP, Kempker RR, Peloquin CA. Population Pharmacokinetics of Linezolid in Tuberculosis Patients: Dosing Regimen Simulation and Target Attainment Analysis. Antimicrob Agents Chemother. 2020 Sep 21;64(10):e01174-20. doi: 10.1128/AAC.01174-20. Print 2020 Sep 21. PMID 32778547
- [Background] Millard J, Pertinez H, Bonnett L, Hodel EM, Dartois V, Johnson JL, Caws M, Tiberi S, Bolhuis M, Alffenaar JC, Davies G, Sloan DJ. Linezolid pharmacokinetics in MDR-TB: a systematic review, meta-analysis and Monte Carlo simulation. J Antimicrob Chemother. 2018 Jul 1;73(7):1755-1762. doi: 10.1093/jac/dky096. PMID 29584861
- [Background] Wasserman S, Brust JCM, Abdelwahab MT, Little F, Denti P, Wiesner L, Gandhi NR, Meintjes G, Maartens G. Linezolid toxicity in patients with drug-resistant tuberculosis: a prospective cohort study. J Antimicrob Chemother. 2022 Mar 31;77(4):1146-1154. doi: 10.1093/jac/dkac019. PMID 35134182
- [Background] Song T, Lee M, Jeon HS, Park Y, Dodd LE, Dartois V, Follman D, Wang J, Cai Y, Goldfeder LC, Olivier KN, Xie Y, Via LE, Cho SN, Barry CE 3rd, Chen RY. Linezolid Trough Concentrations Correlate with Mitochondrial Toxicity-Related Adverse Events in the Treatment of Chronic Extensively Drug-Resistant Tuberculosis. EBioMedicine. 2015 Oct 9;2(11):1627-33. doi: 10.1016/j.ebiom.2015.09.051. eCollection 2015 Nov. PMID 26870788
- [Background] Wasserman S, Denti P, Brust JCM, Abdelwahab M, Hlungulu S, Wiesner L, Norman J, Sirgel FA, Warren RM, Esmail A, Dheda K, Gandhi NR, Meintjes G, Maartens G. Linezolid Pharmacokinetics in South African Patients with Drug-Resistant Tuberculosis and a High Prevalence of HIV Coinfection. Antimicrob Agents Chemother. 2019 Feb 26;63(3):e02164-18. doi: 10.1128/AAC.02164-18. Print 2019 Mar. PMID 30617089
- [Background] Srivastava S, Magombedze G, Koeuth T, Sherman C, Pasipanodya JG, Raj P, Wakeland E, Deshpande D, Gumbo T. Linezolid Dose That Maximizes Sterilizing Effect While Minimizing Toxicity and Resistance Emergence for Tuberculosis. Antimicrob Agents Chemother. 2017 Jul 25;61(8):e00751-17. doi: 10.1128/AAC.00751-17. Print 2017 Aug. PMID 28584143
- [Background] Kamp J, Bolhuis MS, Tiberi S, Akkerman OW, Centis R, de Lange WC, Kosterink JG, van der Werf TS, Migliori GB, Alffenaar JC. Simple strategy to assess linezolid exposure in patients with multi-drug-resistant and extensively-drug-resistant tuberculosis. Int J Antimicrob Agents. 2017 Jun;49(6):688-694. doi: 10.1016/j.ijantimicag.2017.01.017. Epub 2017 Apr 4. PMID 28389352
- [Background] Rao GG, Konicki R, Cattaneo D, Alffenaar JW, Marriott DJE, Neely M; IATDMCT Antimicrobial Scientific Committee. Therapeutic Drug Monitoring Can Improve Linezolid Dosing Regimens in Current Clinical Practice: A Review of Linezolid Pharmacokinetics and Pharmacodynamics. Ther Drug Monit. 2020 Feb;42(1):83-92. doi: 10.1097/FTD.0000000000000710. PMID 31652190
- [Background] Zhou W, Nie W, Wang Q, Shi W, Yang Y, Li Q, Zhu H, Liu Z, Ding Y, Lu Y, Chu N. Linezolid Pharmacokinetics/Pharmacodynamics-Based Optimal Dosing for Multidrug-Resistant Tuberculosis. Int J Antimicrob Agents. 2022 Jun;59(6):106589. doi: 10.1016/j.ijantimicag.2022.106589. Epub 2022 Apr 9. PMID 35405268
- [Background] Cattaneo D, Orlando G, Cozzi V, Cordier L, Baldelli S, Merli S, Fucile S, Gulisano C, Rizzardini G, Clementi E. Linezolid plasma concentrations and occurrence of drug-related haematological toxicity in patients with gram-positive infections. Int J Antimicrob Agents. 2013 Jun;41(6):586-9. doi: 10.1016/j.ijantimicag.2013.02.020. Epub 2013 Apr 4. PMID 23562639
- [Background] Eimer J, Frechet-Jachym M, Le Du D, Caumes E, El-Helali N, Marigot-Outtandy D, Mechai F, Peytavin G, Pourcher V, Rioux C, Yazdanpanah Y, Robert J, Guglielmetti L; LZDM group. Association Between Increased Linezolid Plasma Concentrations and the Development of Severe Toxicity in Multidrug-Resistant Tuberculosis Treatment. Clin Infect Dis. 2023 Feb 8;76(3):e947-e956. doi: 10.1093/cid/ciac485. PMID 35717636
- [Background] Mase A, Lowenthal P, True L, Henry L, Barry P, Flood J. Low-Dose Linezolid for Treatment of Patients With Multidrug-Resistant Tuberculosis. Open Forum Infect Dis. 2022 Oct 5;9(12):ofac500. doi: 10.1093/ofid/ofac500. eCollection 2022 Dec. PMID 36601556
- [Background] Begg EJ, Barclay ML, Kirkpatrick CJ. The therapeutic monitoring of antimicrobial agents. Br J Clin Pharmacol. 1999 Jan;47(1):23-30. doi: 10.1046/j.1365-2125.1999.00850.x. PMID 10073735
- [Background] Haley CA, Schechter MC, Ashkin D, Peloquin CA, Peter Cegielski J, Andrino BB, Burgos M, Caloia LA, Chen L, Colon-Semidey A, DeSilva MB, Dhanireddy S, Dorman SE, Dworkin FF, Hammond-Epstein H, Easton AV, Gaensbauer JT, Ghassemieh B, Gomez ME, Horne D, Jasuja S, Jones BA, Kaplan LJ, Khan AE, Kracen E, Labuda S, Landers KM, Lardizabal AA, Lasley MT, Letzer DM, Lopes VK, Lubelchek RJ, Patricia Macias C, Mihalyov A, Misch EA, Murray JA, Narita M, Nilsen DM, Ninneman MJ, Ogawa L, Oladele A, Overman M, Ray SM, Ritger KA, Rowlinson MC, Sabuwala N, Schiller TM, Schwartz LE, Spitters C, Thomson DB, Tresgallo RR, Valois P, Goswami ND; BPaL Implementation Group. Implementation of Bedaquiline, Pretomanid, and Linezolid in the United States: Experience Using a Novel All-Oral Treatment Regimen for Treatment of Rifampin-Resistant or Rifampin-Intolerant Tuberculosis Disease. Clin Infect Dis. 2023 Oct 5;77(7):1053-1062. doi: 10.1093/cid/ciad312. PMID 37249079
- [Background] Pea F, Viale P, Cojutti P, Del Pin B, Zamparini E, Furlanut M. Therapeutic drug monitoring may improve safety outcomes of long-term treatment with linezolid in adult patients. J Antimicrob Chemother. 2012 Aug;67(8):2034-42. doi: 10.1093/jac/dks153. Epub 2012 May 2. PMID 22553142
- [Background] Schwartz D, Lellouch J. Explanatory and pragmatic attitudes in therapeutical trials. J Chronic Dis. 1967 Aug;20(8):637-48. doi: 10.1016/0021-9681(67)90041-0. No abstract available. PMID 4860352
- [Background] Ford I, Norrie J. Pragmatic Trials. N Engl J Med. 2016 Aug 4;375(5):454-63. doi: 10.1056/NEJMra1510059. No abstract available. PMID 27518663
- [Background] UNAIDS. Global AIDS Update. Geneva 2023.
- [Background] Brust JC, Shah NS, Scott M, Chaiyachati K, Lygizos M, van der Merwe TL, Bamber S, Radebe Z, Loveday M, Moll AP, Margot B, Lalloo UG, Friedland GH, Gandhi NR. Integrated, home-based treatment for MDR-TB and HIV in rural South Africa: an alternate model of care. Int J Tuberc Lung Dis. 2012 Aug;16(8):998-1004. doi: 10.5588/ijtld.11.0713. Epub 2012 Jun 5. PMID 22668560
- [Background] Loveday M, Wallengren K, Voce A, Margot B, Reddy T, Master I, Brust J, Chaiyachati K, Padayatchi N. Comparing early treatment outcomes of MDR-TB in decentralised and centralised settings in KwaZulu-Natal, South Africa. Int J Tuberc Lung Dis. 2012 Feb;16(2):209-15. doi: 10.5588/ijtld.11.0401. PMID 22236922
- [Background] Department of Health South Africa. Interim clinical guidance for the implementation of injectable-free regimens for rifampicin-resistant tuberculosis in adults, adolescents and children. 2018.
- [Background] Medecins Sans Frontieres. South Africa Becomes First Country to Include New, More Effective DR-TB Drug in Standard Treatment https://wwwdoctorswithoutbordersorg/latest/south-africa-becomes-first-country-include-new-more-effective-dr-tb-drug-standard-treatment (accessed August 9, 2023) 2018.
- [Background] Ndjeka N, Conradie F, Schnippel K, Hughes J, Bantubani N, Ferreira H, Maartens G, Mametja D, Meintjes G, Padanilam X, Variava E, Pym A, Pillay Y. Treatment of drug-resistant tuberculosis with bedaquiline in a high HIV prevalence setting: an interim cohort analysis. Int J Tuberc Lung Dis. 2015 Aug;19(8):979-85. doi: 10.5588/ijtld.14.0944. PMID 26162365
- [Background] U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS. Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1. [July 2017]. Available from: https://rsc.niaid.nih.gov/sites/default/files/daidsgradingcorrectedv21.pdf (accessed Sep 10, 2023).
- [Background] McArthur JH. The reliability and validity of the subjective peripheral neuropathy screen. J Assoc Nurses AIDS Care. 1998 Jul-Aug;9(4):84-94. doi: 10.1016/S1055-3290(98)80048-4. PMID 9658364
- [Background] Cherry CL, Wesselingh SL, Lal L, McArthur JC. Evaluation of a clinical screening tool for HIV-associated sensory neuropathies. Neurology. 2005 Dec 13;65(11):1778-81. doi: 10.1212/01.wnl.0000187119.33075.41. PMID 16344522
- [Background] Rusch-Gerdes S, Pfyffer GE, Casal M, Chadwick M, Siddiqi S. Multicenter laboratory validation of the BACTEC MGIT 960 technique for testing susceptibilities of Mycobacterium tuberculosis to classical second-line drugs and newer antimicrobials. J Clin Microbiol. 2006 Mar;44(3):688-92. doi: 10.1128/JCM.44.3.688-692.2006. PMID 16517840
- [Background] World Health Organization. Definitions and reporting framework for tuberculosis - 2013 revision (updated December 2014 and January 2020). WHO/HTM/TB/20132 Geneva.
- [Background] Boak LM, Rayner CR, Grayson ML, Paterson DL, Spelman D, Khumra S, Capitano B, Forrest A, Li J, Nation RL, Bulitta JB. Clinical population pharmacokinetics and toxicodynamics of linezolid. Antimicrob Agents Chemother. 2014;58(4):2334-43. doi: 10.1128/AAC.01885-13. Epub 2014 Feb 10. PMID 24514086
- [Background] Friberg LE, Henningsson A, Maas H, Nguyen L, Karlsson MO. Model of chemotherapy-induced myelosuppression with parameter consistency across drugs. J Clin Oncol. 2002 Dec 15;20(24):4713-21. doi: 10.1200/JCO.2002.02.140. PMID 12488418
- [Background] Sharma A, Jusko WJ. Characteristics of indirect pharmacodynamic models and applications to clinical drug responses. Br J Clin Pharmacol. 1998 Mar;45(3):229-39. doi: 10.1046/j.1365-2125.1998.00676.x. PMID 9517366
- [Background] Abdelwahab MT, Wasserman S, Brust JCM, Dheda K, Wiesner L, Gandhi NR, Warren RM, Sirgel FA, Meintjes G, Maartens G, Denti P. Linezolid Population Pharmacokinetics in South African Adults with Drug-Resistant Tuberculosis. Antimicrob Agents Chemother. 2021 Nov 17;65(12):e0138121. doi: 10.1128/AAC.01381-21. Epub 2021 Sep 20. PMID 34543098
- [Background] Bigelow KM, Deitchman AN, Li SY, Barnes-Boyle K, Tyagi S, Soni H, Dooley KE, Savic RM, Nuermberger EL. Pharmacodynamic Correlates of Linezolid Activity and Toxicity in Murine Models of Tuberculosis. J Infect Dis. 2021 Jun 4;223(11):1855-1864. doi: 10.1093/infdis/jiaa016. PMID 31993638
- [Background] Stalker DJ, Jungbluth GL. Clinical pharmacokinetics of linezolid, a novel oxazolidinone antibacterial. Clin Pharmacokinet. 2003;42(13):1129-40. doi: 10.2165/00003088-200342130-00004. PMID 14531724
- [Background] Svensson EM, Aweeka F, Park JG, Marzan F, Dooley KE, Karlsson MO. Model-based estimates of the effects of efavirenz on bedaquiline pharmacokinetics and suggested dose adjustments for patients coinfected with HIV and tuberculosis. Antimicrob Agents Chemother. 2013 Jun;57(6):2780-7. doi: 10.1128/AAC.00191-13. Epub 2013 Apr 9. PMID 23571542
- [Background] Falzon D, Gandhi N, Migliori GB, Sotgiu G, Cox HS, Holtz TH, Hollm-Delgado MG, Keshavjee S, DeRiemer K, Centis R, D'Ambrosio L, Lange CG, Bauer M, Menzies D; Collaborative Group for Meta-Analysis of Individual Patient Data in MDR-TB. Resistance to fluoroquinolones and second-line injectable drugs: impact on multidrug-resistant TB outcomes. Eur Respir J. 2013 Jul;42(1):156-68. doi: 10.1183/09031936.00134712. Epub 2012 Oct 25. PMID 23100499